CLINICAL TRIAL: NCT04790084
Title: Changes of Three-dimensional Choroidal Vascular Index by Optical Coherence Tomography in Common Fundus Diseases
Brief Title: Three-dimensional Choroidal Vascularity Index in Common Fundus Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Changzheng Chen, Chief of Department of Ophthalmology, Renmin Hospital of Wuhan University
Other Study IDs: 3DCVICFD
Record Dates: First submitted 2021-03-03; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Choroid
Keywords: choroidal vascularity index; fundus disease; choroidal blood flow

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Healthy-Myopia-CSC: Cross-sectional study, no intervention, only collecting OCT,OCTA images and other eye parameters of patients.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Explore the changes of choroidal blood perfusion in common fundus diseases by three-dimensional choroidal vascularity index, an optical coherence tomography (OCT) parameter.

DETAILED DESCRIPTION:
Compared with the choroidal vascularity index on a single OCT image, the three-dimensional choroidal vascularity index can evaluate the choroidal changes of chorioretinal diseases as a whole. In this study, the choroidal changes of patients with common fundus diseases were systematically evaluated by collecting OCT and optical coherence tomography angiography (OCTA) images of patients with common fundus diseases, especially in healthy people, myopic people and patients with central serous chorioretinopathy.

ELIGIBILITY:
1. Healthy participants (1) Inclusion Criteria: 1) without systemic diseases such as diabetes and hypertension 2) best corrected visual acuity BCVA ≥ 1.0 3) aged 18 years or older (2) Exclusion criteria: 1) equivalent spherical refraction between -3 diopters and + 1.0 diopters 2) any visible lesions in the retina, optic nerve, or choroid 3) history of refractive or intraocular surgery
2. Myopia group (1) Inclusion Criteria: 1) equivalent spherical refraction greater than -0.25 diopters 2) without systemic diseases such as diabetes and hypertension 3) Best corrected visual acuity (BCVA) ≥ 1.0 4) aged 10 years or older (2) Exclusion criteria: 1) history of refractive or intraocular surgery 2) history of laser therapy 3) other systemic diseases that may affect the choroid
3. Central serous chorioretinopathy (CSC) group (1) Inclusion Criteria: 1) a diagnosis of CSC (2) Exclusion criteria: 1) high myopia or hyperopia (greater than 26 or +3 diopters of refractive error) 3) other systemic diseases that may affect the choroid 4) any other associated retinal pathology 5) history of refractive or intraocular surgery

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Chinese
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2024-03-10 (Estimated); Study Completion 2024-03-10 (Estimated)

PRIMARY OUTCOMES:
Three-dimensional choroidal vascularity index | baseline, pre-intervention
  Three-dimensional choroidal vascularity index of healthy people and patients with common fundus diseases, based on optical coherence tomography.

SECONDARY OUTCOMES:
Choriocapillaris flow deficits% | baseline, pre-intervention
  Choriocapillaris flow deficits% of healthy people and patients with common fundus diseases, based on optical coherence tomography angiography.

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China